CLINICAL TRIAL: NCT01378104
Title: The Response of Reducing Dose of Peginterferon Alfa-2a in Koreans With Chronic Hepatitis C Genotype 1; Randomized Controlled Multicenter Study 100% Versus 80%
Brief Title: 100% VS 80% Of Pegasys In Koreans With Chronic Hepatitis C (CHC)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The Catholic University of Korea (Other)
Collaborators: Ulsan University Hospital (Other); National Health Insurance Service Ilsan Hospital (Other); Inje University (Other); Soonchunhyang University Hospital (Other); Yonsei University (Other); Chungnam National University (Other); Keimyung University (Other); Kyungpook National University Hospital (Other); Konyang University Hospital (Other); Inha University Hospital (Other); Hallym University Medical Center (Other)
Responsible Party: Principal Investigator, Jung Hyun Kwon, Assistant professor, The Catholic University of Korea
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PEGASYS100:80
Record Dates: First submitted 2011-06-16; First posted 2011-06-22 (Estimated); Results first posted 2013-03-08 (Estimated); Last update posted 2013-03-08 (Estimated); Status verified 2013-02

CONDITIONS: Sustained Virologic Response; IL28B Polymorphism
Keywords: reducing dose of peginterferon; chronic hepatitis c; Koreans; IL28B polymorphism
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — peginterferon alfa-2a

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 80% dosage group of peginterferon alfa 2a (Experimental): This group patients will treated the same full dose (180ug/week) of peginterferon alfa 2a during the first 12 weeks and then reduce the 75% dose (135ug/week) of peginterferon alfa 2a during remnant 36 weeks. At a result, these patients treated with 80% dosage of originally prescribed peginterferon alfa-2a for standard 48 weeks of treatment.
  Interventions: Drug: peginterferon alfa 2a (pegasys)
- 100% dosage group of peginterferon alfa 2a (Active Comparator): These group patients would be treated with standard dose 180 ug/week for 48 weeks.
  Interventions: Drug: peginterferon alfa-2a (pegasys)

INTERVENTIONS:
Drug: peginterferon alfa 2a (pegasys) — dosage form; 180ug/week during first 12 weeks and then 135 ug/week during 36 weeks otherwise unremarkable
  Other Names: Roche
  Arms: 80% dosage group of peginterferon alfa 2a
Drug: peginterferon alfa-2a (pegasys) — These patients would be treated with standard dose 180ug /week for 48 weeks. In general, the patient with CHC genotype 1is guided with treatment with pegasys 180ug /week and ribavirin 1000-1200 mg/day for 48 weeks. We do not make intervention of ribavirin dose.
  Other Names: Roche
  Arms: 100% dosage group of peginterferon alfa 2a

SUMMARY:
1. Randomized controlled multicenter study
2. The response of reducing dose of peginterferon alfa-2a in Koreans with chronic hepatitis C genotype 1
3. IL28B polymorphism in Koreans with CHC

DETAILED DESCRIPTION:
The virologic response of Koreans to combination therapy for chronic hepatitis C is similar to non-Asians; however, dose modification occurs more frequently in Koreans.

-When we evaluated the rates of peginterferon α-2a and ribavirin dose modifications and their effect on the virologic response in Koreans, we suggested that using at least 80% of the peginterferon α-2a dose in Koreans not only maintains SVR but also reduces drug side effects during the entire treatment period and a lower dose of ribavirin may be as efficacious as a standard dose(Korean J Intern Med 2009;24:203-211).

So we investigate whether the group of 80% use dosage of peginterferon alfa-2a did not show inferior response rather than that of 100 % use dosage group and minimize the adverse events.

There are recently reports that Koreans have favorable IL28B SNP for CHC treatment.

-We investigate the IL28B polymorphism in Koreans with CHC and this result can effect on the SVR depending on the dosage of peginterferon alfa 2a

ELIGIBILITY:
Inclusion Criteria:

* chronic hepatitis C (anti HCV+, HCV RNA +)
* Genotype 1
* over 18 year-old
* Pregnancy test negative if women of childbearing age

Exclusion Criteria:

* pregnant women or breast feeding women
* systemic chemotherapy or steroid therapy before 6 months of trial
* Coinfection with HAV, HBV, and HIV
* Other liver disease such as hemochromatosis, autoimmune hepatitis, metabolic liver disease, alcoholic liver disease, toxic hepatitis
* Hepatocellular carcinoma
* Evidence of decompensation such as variceal bleeding,ascites, encephalopathy
* ANC less than 1500, platelet less than 90k
* Cr more than 1.5 of UNL
* Severe psychiatric problem
* Poorly controlled thyroid disease
* Severe retinopathy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 178 (Actual)
Dates: Start 2008-10; Primary Completion 2011-09 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jung Hyun Kwon, MD, Assistant professor, Principal Investigator — The Catholic University of Korea
Locations (14):
- South Korea (14):
  - Soonchunghyang University Hospital, Bucheon-si
  - Hallym University Chunchun Medical center, Chunchun
  - Keimyung University hospital, Daegu
  - Kyungpook National University Hospital, Daegu
  - Ghungnam National University hospital, Daejun
  - Konyang University hospital, Daejun
  - Incheon St. Mary's Hospital, Incheon
  - Inha University hospital, Incheon
  - Inje University, Ilsan Paik Hospital, Koyang-si
  - NHIC Ilsan hospital, Koyang-si
  - Inje University, Pusan Paik Hospital, Pusan
  - Seoul St. Mary's Hospital, The Catholic University of Korea, Seoul
  - Ulsan university, Ulsan
  - Yonsei University, Wonju Hospital, Wŏnju

RESULTS

PARTICIPANT FLOW:
Recruitment Details: enrollment date : 2009-2011 recruitment period : 2009-2012 type location: 14 university hospital
Pre-assignment Details: no excluded patients before assignment to groups
Groups:
- 100% Dosage Group of Peginterferon Alfa 2a: These group patients would be treated with standard dose 180 ug/week for 48 weeks.
  peginterferon alfa-2a (pegasys) : These patients would be treated with standard dose 180ug /week for 48 weeks.
  In general, the patient with CHC genotype 1is guided with treatment with pegasys 180ug /week and ribavirin 1000-1200 mg/day for 48 weeks. We do not make intervention of ribavirin dose.
- 80% Dosage Group of Peginterferon Alfa 2a: This group patients will treated the same full dose (180ug/week) of peginterferon alfa 2a during the first 12 weeks and then reduce the 75% dose (135ug/week) of peginterferon alfa 2a during remnant 36 weeks. At a result, these patients treated with 80% dosage of originally prescribed peginterferon alfa-2a for standard 48 weeks of treatment.
  peginterferon alfa 2a (pegasys) : dosage form; 180ug/week during first 12 weeks and then 135 ug/week during 36 weeks otherwise unremarkable
Period: Overall Study
Arm/Group | 100% Dosage Group of Peginterferon Alfa 2a | 80% Dosage Group of Peginterferon Alfa 2a
Started | 92 | 86
Completed | 65 | 60
Not Completed | 27 | 26
Not completed — Adverse Event | 8 | 8
Not completed — Lack of Efficacy | 7 | 5
Not completed — Withdrawal by Subject | 12 | 13

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 100% Dosage Group of Peginterferon Alfa 2a | 80% Dosage Group of Peginterferon Alfa 2a | Total
Number analyzed (Participants) | 92 | 86 | 178
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 88 | 81 | 169
  >=65 years | 4 | 5 | 9
Age Continuous [Mean (Standard Deviation); unit: years] | 48.5 (10.6) | 48.7 (11.5) | 48.6 (11.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42 | 45 | 87
  Male | 50 | 41 | 91
Region of Enrollment [Number; unit: participants]
  Korea, Republic of | 92 | 86 | 178

OUTCOME MEASURES:

1. Primary Outcome: Sustained Virologic Response Depending on the Dosage of Peginterferon Alfa 2a
Description: We investigate whether the SVR between 100% and 80% group of peginterferon alfa 2a is not different.
Time Frame: post treatment 24 weeks
Population: We present the result of intention-to-treat analysis.
Measure: Number; unit: participants who achieved SVR
Arm/Group | 100% Dosage Group of Peginterferon Alfa 2a | 80% Dosage Group of Peginterferon Alfa 2a
Number analyzed (Participants) | 92 | 86
participants who achieved SVR | 52 | 44

2. Secondary Outcome: IL28B Polymorphism Effect on SVR
Description: We additionally investigate the IL28B polymorphism and this result can effect on the SVR depending on dosage of peginterferon alfa-2a.
Time Frame: post treatment 24 weeks
Population: The patients who agreed to check the genotype were analysed.
Measure: Number; unit: percentage of SVR
Groups:
- Favourable IL28B Genotype: These group patients show the IL28B rs12979860CC and rs8099917TT.
- The Patients With Unfavourable IL28B Genotype: These group patients show the IL28B rs12979860 CT or TT and rs8099917 TG or GG.
Arm/Group | Favourable IL28B Genotype | The Patients With Unfavourable IL28B Genotype
Number analyzed (Participants) | 82 | 18
percentage of SVR | 71.9 | 33.3

ADVERSE EVENTS:
Arm/Group | 100% Dosage Group of Peginterferon Alfa 2a | 80% Dosage Group of Peginterferon Alfa 2a
Serious Adverse Events (participants affected / at risk) | 0/92 | 0/86
Other Adverse Events (participants affected / at risk) | 45/92 | 49/86
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 100% Dosage Group of Peginterferon Alfa 2a (N=92) | 80% Dosage Group of Peginterferon Alfa 2a (N=86)
laboratory adverse events (Blood and lymphatic system disorders) | 45 (54) | 49 (49) — Neutropenia, thrombocytopenia, anemia

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No